CLINICAL TRIAL: NCT05767021
Title: A Multicenter, Phase 3b, Open-Label, Single-Arm Study to Investigate Bowel Urgency and Its Relationship With Other Outcome Measures in Adults With Moderately to Severely Active Ulcerative Colitis Treated With Mirikizumab
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: LUCENT-URGE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18551; I6T-MC-AMBZ (Other: Eli Lilly and Company); 2022-502393-16-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-02-08; First posted 2023-03-14 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 300 mg Mirikizumab (Experimental): Participants received 300 milligram (mg) mirikizumab every 4 weeks (Q4W) at week 0, 4, and 8 administered intravenously (IV).
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
Drug: Mirikizumab — Administered Subcutaneously (SC)
  Other Names: LY3074828

SUMMARY:
A study to investigate bowel urgency in adults with moderately to severely active ulcerative colitis (UC) treated with mirikizumab. The study will have 4 periods and will last for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have an established diagnosis of UC for ≥3 months
* Have confirmed diagnosis of moderately for severely active UC
* Have current bowel urgency
* Have demonstrated an inadequate response to, a loss of response to, or an intolerance to conventional or to biologic/Janus Kinase (JAK) inhibitor/sphingosine-1-phosphate (S1P) receptor modulator therapy for UC.

Exclusion Criteria:

* Have Crohn's disease (CD)
* Have inflammatory bowel disease-unclassified, formerly known as indeterminate colitis, or
* Have ulcerative proctitis, disease limited to the rectum, that is, distal to the recto-sigmoid junction, which lies approximately 10 to 15 centimeter (cm) from anal verge.
* Have an inherited immunodeficiency syndrome or a monogenic cause of UC-like colonic inflammation
* Have any history or current evidence of cancer of the gastrointestinal tract
* Have active tuberculosis
* Have HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (120):
- United States (49):
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Om Research, LLC, Lancaster, California
  - California Medical Research Associates, Inc., Northridge, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Central Florida Gastro Research, Clearwater, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Research Associates of South Florida, Miami, Florida
  - Advanced Research Associates, LLC, Miami, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - International Center for Research LLC, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - IU Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, New Albany, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - GI Alliance/ Metairie, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - NY Scientific, Brooklyn, New York
  - Digestive Health Partners - Research Department, Asheville, North Carolina
  - Charlotte Gastroenterolgy & Hepatology, Charlotte, North Carolina
  - Innovo Research:Wilmington Health, Wilmington, North Carolina
  - Optimed Research, LTD, Columbus, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Cordova, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Clinical Trial Network, Houston, Texas
  - Houston Endoscopy And Research Center, LLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Citrine Institute for Research and Wellness, Katy, Texas
  - AngioCardiac Care of Texas, PA, McAllen, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Gastroenterology Associates of Texas - Denise Rodriguez, Sugar Land, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - GI Alliance Research Webster, Webster, Texas
  - Care Access Research - Ogden, Ogden, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Washington Gastroenterology dba GI Alliance, Tacoma, Washington
- Belgium (2):
  - Universitair Ziekenhuis Gent - Gastro IBD, Ghent
  - UZ Leuven - E507 Studies IBD tav Tine Hermans, Leuven
- Czechia (7):
  - Vojenska nemocnice Brno, Interni oddeleni, Brno, Czech Republic
  - GastroJeka s.r.o, Klatovy, Czech Republic
  - FN Ostrava, Interní Klinika, Ostrava, Czech Republic
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové, Hradec Králové
  - MUDr. Gregar, s.r.o., Olomouc, Olomoucký kraj
  - SurGal clinic s.r.o., Brno
  - PreventaMed, s.r.o., Olomouc
- France (13):
  - Hospices Civils de Lyon - Hôpital Lyon Sud - ARC HGE bâtiment 3I, Lyon - Pierre Benite, France
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - CHU Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques
  - Chu Besancon, Besançon
  - CHU de LILLE - Bureau des ARCs Gastro - HPDD, Lille
  - Hôpital Saint-Eloi Pôle Digestif ,APEMAD - Recherche clinique, Montpellier
  - CHU Nantes, Nantes
  - Clinique Jules Verne, Nantes
  - Unité de Recherche Clinique (4èmeB), Nice
  - Chu de Reims - Hôpital Robert Debré, Reims
  - CHU de Saint-Etienne, Saint-Etienne
  - Chru Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (3):
  - Praxis Dr. M. Mross - Gastroenterologie, Berlin
  - DRK Kliniken Berlin Westend, Gastroenterologie, Studienbüro, Berlin
  - Universitätsklinikum Leipzig, Med. Klinik II, Leipzig
- Hungary (5):
  - Bugat Pal Korhaz, Gyöngyös, Heves County
  - Clinepert kft, Budapest
  - Semmelweis Egyetem, Belgyógyászati es Hematológiai Klinika, Budapest
  - Pannónia Magánorvosi Centrum, Budapest
  - Clinfan Ltd. Gastroenterology Clinic, Szekszárd
- Italy (8):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - IRCCS Saverio de Bellis, National Institute of Gastroenterology, Castellana Grotte
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - Irccs Ospedale San Raffaele, Gastroenterologia/Ibd Unit, Settore G Piano -1, Milan
  - Fondazione Policlinico Agostino Gemelli IRCCS_ CEMAD, Roma
  - Uoc Gastroenterologia - Policlinico Tor Vergata, Roma
  - IRCCS Istituto Clinico Humanitas- Centro Malattie Infiammatorie Intestinali, Rozzano
  - A.O.Ordine Mauriziano, SC Gastroenterologia, ambulatorio endoscopia digestiva, Torino
- Poland (23):
  - Solumed Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - MZ Badania Słowik Zymła Sp.j., Knurów, Silesian Voivodeship
  - Centrum Medyczne Medyk, Rzeszów, Subcarpathian
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Vitamed Galaj I Cichomski sp.j., Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - KRAKOWSKIE CENTRUM MEDYCZNE Sp. z o.o, Krakow
  - Topolowa Medicenter Ryszawa & Wspólnicy Sp.j., Krakow
  - IP Clinic, Lodz
  - Med-GASTR SP. Z O.O., SP.K., Lodz
  - AmiCare Sp. z o.o. Sp. K., Lodz
  - Bonifraterskie Centrum Medyczne sp. z o.o, Lodz
  - Allmedica Badania Kliniczne Sp. z o.o. Sp. k., Nowy Targ
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - Nowe Zdrowie-Ck, Kiełtucki I Wspólnicy Sp. J., Staszów
  - DC-MED Sp. z o.o. s.k., Swidnica
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - NZOZ FOR MED sp. z o.o., Wadowice
  - FutureMeds sp. z o. o., Wroclaw
  - PlanetMed Sp.z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Centrum Medyczne Kuba Med 2 Sp. z o.o. ETG Zamosc, Zamość
- Slovakia (7):
  - Fakultná nemocnica s poliklinikou F. D. Roosevelta Banská Bystrica gastroenterologická ambulancia, II. Interná klinika SZU, Banská Bystrica, Slovak Republic
  - ALIAN s.r.o., Bardejov, Slovak Republic
  - CLINIQ, s.r.o, Bratislava, Slovak Republic
  - GASTRO AMBULANCIA, poliklinika Ťahanovce, Košice, Slovak Republic
  - Fakultna nemocnica Nitra, Interna klinika, Nitra, Slovak Republic
  - KM Management, spol. s.r.o, Nitra Stare Mesto, Slovak Republic
  - Accout Center s.r.o., Šahy, Slovak Republic
- United Kingdom (3):
  - Fairfield General Hospital, Bury, Great Britain
  - Clinical Research Unit, Royal Liverpool University Hospital, Waltham, Waltham Forest
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Time Frame:
  Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Mirikizumab (LY3074828) in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT-URGE) — https://trials.lilly.com/en-US/trial/394020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Current results reporting analysis is only for the primary outcome data per Primary completion date (August 9, 2024) and final results will be presented at the time of reporting the final results, i.e., no later than September 2026.
Period: Overall Study
Arm/Group | 300 mg Mirikizumab
Started | 172
Received at Least One Dose of Study Drug | 172
Completed (This Period includes all participants who completed the study for 12-weeks treatment period.) | 155
Not Completed | 17
Not completed — Adverse Event | 2
Not completed — Protocol Deviation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 11
Not completed — Assigned Treatment by Mistake | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 300 mg Mirikizumab: Participants received 300 mg mirikizumab Q4W at week 0, 4, and 8 administered IV.
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.10 (14.352)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 151
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 150
  More than one race | 1
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 7
  United States | 33
  Czechia | 18
  Poland | 50
  Italy | 32
  United Kingdom | 6
  Slovakia | 10
  France | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bowel Urgency Severity Urgency Numeric Rating Scale (UNRS)
Description: The UNRS is a single participant reported item that measures the severity for the urgency (sudden or immediate need) to have a bowel movement in the past 24 hours using an 11-point NRS ranging from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicate more severe urgency.
  Baseline Observation Carried Forward (BOCF) endpoint was defined as the baseline value for participants discontinued during acute phase and defined as the last non-missing observation in the treatment phase for all other randomized participants.
Time Frame: Baseline, Week 12
Population: All enrolled participants who received at least one dose of study drug (regardless of whether the participant does not receive the correct treatment or otherwise does not follow the protocol) with a non-missing baseline and BOCF endpoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
score on a scale | -3.25 [-3.63 to -2.87]

2. Secondary Outcome: Change From Baseline in Bowel Urgency Frequency (BUF)
Description: BUF is participant reported single item measure of the number of urgent bowel movements reported in the past 24 hours.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: counts of urgent bowel movements/day
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
counts of urgent bowel movements/day | -3.83 [-4.33 to -3.33]

3. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Improvement in BUF
Description: This outcome measures the percentage of participants who experience a clinically meaningful reduction in the frequency of bowel urgency episodes from baseline to the 12 week treatment period. Results for this outcome will be reported during final results posting.
Time Frame: Baseline to Week 12
Reporting Status: Not Posted, anticipated posting 2026-09

4. Secondary Outcome: Percentage of Participants With Stool Deferral Time (SDT) Intervals at Week 12
Description: The SDT is a participant-reported single item measure of the average duration a patient could delay defecation in the past 24 hours. The shortest weekly SDT is used for analysis of SDT in minutes by taking the shortest response (i.e. minimum value) available over the past 7 days, where no urgency is treated as the largest value. The SDT categories were:<1 min, ≥1 min to <2 min, ≥2 min to <5 min, ≥5 min to <15 min, and ≥15 min or no urgency. No urgency indicates participant's selected "Did not feel urge to have a bowel movement in the past 24 hours" for all available days in 7-day period.
Time Frame: Week 12
Population: All enrolled participants who received at least one dose of study drug (regardless of whether the participant does not receive the correct treatment or otherwise does not follow the protocol)
Measure: Number; unit: percentage of participants
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
percentage of participants
  <1 min | 8.7
  >=1 to <2 min | 21.5
  >=2 to <5 min | 30.2
  >=5 to <15 min | 23.8
  >=15 min or no urgency | 15.7

5. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Improvement of SDT
Description: This outcome measures the percentage of participants who demonstrate a clinically meaningful improvement in SDT. Results for this outcome will be reported during final results posting.
Time Frame: Week 12
Reporting Status: Not Posted, anticipated posting 2026-09

6. Secondary Outcome: Percentage of Participants Achieving Both Clinical Remission, Based on the Modified Mayo Score (MMS) and a Rounded Urgency Numeric Rating Scale (UNRS) Score of ≤1
Description: Clinical remission based on MMS is defined as Stool Frequency (SF) sub score (range 0-3, higher is worse) = 0, or SF = 1 with a ≥1- point decrease from baseline, and
  1. Rectal Bleeding (RB) sub score (range 0-3, higher is worse) = 0, and
  2. Endoscopic sub score (ES) (range 0-3, higher is worse) = 0 or 1 (excluding friability).
  UNRS measures bowel urgency severity (range 0 to 10; Higher scores indicate more severe urgency)
  This outcome assesses the proportion of participants who achieved both a clinical response, as defined by an MMS, and an improvement of ≥3 points from baseline in a UNRS score at Week 12.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
percentage of participants | 5.23

7. Secondary Outcome: Percentage of Participants Achieving Both Clinical Response, Based on the Modified Mayo Score (MMS) and a Rounded Urgency Numeric Rating Scale (UNRS) Score ≥3 Points of Improvement From Baseline
Description: Clinical response based on MMS is defined as:
  1. A change in the MMS of ≤ -2 points and ≤ -30% change from baseline, and
  2. A change of ≤-1 point in the RB subscore (range 0-3, higher is worse) from baseline or a RB score of 0 or 1.
  UNRS measures bowel urgency severity (range 0 to 10; Higher scores indicate more severe urgency)
  This outcome measures the percentage of participants achieving both, clinical response, based on the MMS, and a UNRS score of ≥3 points of improvement from baseline at 12 weeks.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 172
percentage of participants | 44.19

8. Secondary Outcome: Pairwise Correlations Between the Urgency Numeric Rating Scale (UNRS), Baseline in Bowel Urgency Frequency (BUF), Stool Deferral Time (SDT) and Absorbent Product Use (APU) Measures
Description: UNRS measures bowel urgency severity (range 0 to 10; Higher scores indicate more severe urgency).
  BUF measures the number of urgent bowel movements reported in the past 24 hours.
  SDT measures the average duration a patient could delay defecation in the past 24 hours.
  APU is a single item to assess participant's need to wear an adult diaper, pad or protection because of bowel urgency.
  This outcome evaluates the pairwise correlations among four bowel urgency-related measures above.
Time Frame: Baseline to Week 12
Population: All enrolled participants who received at least one dose of study drug and had evaluable data for this outcome (regardless of whether the participant does not receive the correct treatment or otherwise does not follow the protocol).
Measure: Number (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 160
Spearman Correlation Coefficient
  Correlation between UNRS and BUF | 0.68 [0.58 to 0.75]
  Correlation between UNRS and SDT | -0.50 [-0.61 to -0.37]
  Correlation between UNRS and APU: number analyzed (Participants) | 153
  Correlation between UNRS and APU | 0.37 [0.22 to 0.50]
  Correlation between BUF and SDT | -0.47 [-0.58 to -0.34]
  Correlation between BUF and APU: number analyzed (Participants) | 153
  Correlation between BUF and APU | 0.45 [0.31 to 0.56]
  Correlation between SDT and APU: number analyzed (Participants) | 155
  Correlation between SDT and APU | -0.37 [-0.49 to -0.22]

9. Secondary Outcome: Pairwise Correlations Between Change From Baseline in Urgency Numeric Rating Scale (UNRS), Baseline in Bowel Urgency Frequency (BUF), Stool Deferral Time (SDT) and Absorbent Product Use (APU) Measures
Description: UNRS measures bowel urgency severity (range 0 to 10; Higher scores indicate more severe urgency).
  BUF measures the number of urgent bowel movements reported in the past 24 hours.
  SDT measures the average duration a patient could delay defecation in the past 24 hours.
  APU is a single item to assess participant's need to wear an adult diaper, pad or protection because of bowel urgency.
  This outcome evaluates the pairwise correlations between the change in correlations among four bowel urgency-related measures above.
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 160
Spearman Correlation Coefficient
  Correlation between UNRS and BUF | 0.49 [0.36 to 0.60]
  Correlation between UNRS and SDT | -0.48 [-0.59 to -0.35]
  Correlation between UNRS and APU: number analyzed (Participants) | 150
  Correlation between UNRS and APU | 0.17 [0.01 to 0.32]
  Correlation between BUF and SDT | -0.27 [-0.41 to -0.12]
  Correlation between BUF and APU: number analyzed (Participants) | 150
  Correlation between BUF and APU | 0.16 [0.00 to 0.31]
  Correlation between SDT and APU: number analyzed (Participants) | 152
  Correlation between SDT and APU | 0.07 [-0.09 to 0.23]

10. Secondary Outcome: Correlation Between Urgency Numeric Rating Scale (UNRS), Baseline in Bowel Urgency Frequency (BUF),Stool Deferral Time (SDT) and Absorbent Product Use (APU) Measures,With Quality of Life (QoL)/Functional Outcome Measures and UC Symptom Measures
Description: This outcome evaluates correlations between UNRS, BUF, SDT, APU, and patient-reported outcomes (PROs) related to quality of life (QoL), functional outcomes, and UC symptoms. QoL is assessed using the Inflammatory Bowel Disease Questionnaire (IBDQ), a 32-item patient-completed tool with four domains: bowel (score range 10-70), systemic (5-35), emotional (12-84), and social (5-35). Each item is rated on a 7-point Likert scale (1 = very severe problem,7 = not a problem at all); The total IBDQ score is calculated by summing the scores from all four domains and total score range is 32-224 (Higher = better QoL). Functional outcomes measures: Work Productivity and Activity Impairment (WPAI) questionnaire (four scores derived: absenteeism, presenteeism, productivity loss, activity impairment; each score 0-100%, higher = greater impairment) and Generalized Anxiety Disorder-7 (GAD-7; total score range 0-21, higher = more severe anxiety)... (Continued below due to character constraint)
Time Frame: Baseline to Week 12 UC symptom measures:Patient Global Rating of Severity (PGR-S)(1-6),Patient Global Impression of Change (PGI-C)(1-7),Mayo SF/RB (0-3),Abdominal pain/fatigue NRS (0-10),nocturnal stool frequency;higher=worse severity for all measures.
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 160
Spearman Correlation Coefficient
  UNRS-IBDQ: IBDQ Total score: number analyzed (Participants) | 142
  UNRS-IBDQ: IBDQ Total score | -0.55 [-0.65 to -0.42]
  UNRS-IBDQ: Bowel symptoms: number analyzed (Participants) | 142
  UNRS-IBDQ: Bowel symptoms | -0.48 [-0.60 to -0.35]
  UNRS-IBDQ: Systemic symptoms: number analyzed (Participants) | 142
  UNRS-IBDQ: Systemic symptoms | -0.50 [-0.61 to -0.37]
  UNRS-IBDQ: Emotional function: number analyzed (Participants) | 142
  UNRS-IBDQ: Emotional function | -0.51 [-0.62 to -0.38]
  UNRS-IBDQ: Social function: number analyzed (Participants) | 142
  UNRS-IBDQ: Social function | -0.49 [-0.61 to -0.36]
  UNRS-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 96
  UNRS-WPAI: Work Productivity Loss Score | 0.40 [0.21 to 0.55]
  UNRS-WPAI: Absenteeism Score: number analyzed (Participants) | 107
  UNRS-WPAI: Absenteeism Score | 0.28 [0.10 to 0.45]
  UNRS-WPAI: Presenteeism Score: number analyzed (Participants) | 96
  UNRS-WPAI: Presenteeism Score | 0.39 [0.21 to 0.55]
  UNRS-WPAI: Activity Impairment Score: number analyzed (Participants) | 150
  UNRS-WPAI: Activity Impairment Score | 0.54 [0.41 to 0.64]
  UNRS-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 150
  UNRS-Generalize Anxiety Disorder-7 Score | 0.36 [0.21 to 0.49]
  BUF-IBDQ: IBDQ Total score: number analyzed (Participants) | 142
  BUF-IBDQ: IBDQ Total score | -0.60 [-0.69 to -0.48]
  BUF-IBDQ: Bowel symptoms: number analyzed (Participants) | 142
  BUF-IBDQ: Bowel symptoms | -0.57 [-0.67 to -0.45]
  BUF-IBDQ: Systemic symptoms: number analyzed (Participants) | 142
  BUF-IBDQ: Systemic symptoms | -0.57 [-0.67 to -0.45]
  BUF-IBDQ: Emotional function: number analyzed (Participants) | 142
  BUF-IBDQ: Emotional function | -0.51 [-0.62 to -0.37]
  BUF-IBDQ: Social function: number analyzed (Participants) | 142
  BUF-IBDQ: Social function | -0.58 [-0.68 to -0.46]
  BUF-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 96
  BUF-WPAI: Work Productivity Loss Score | 0.50 [0.33 to 0.63]
  BUF-WPAI: Absenteeism Score: number analyzed (Participants) | 107
  BUF-WPAI: Absenteeism Score | 0.27 [0.08 to 0.43]
  BUF-WPAI: Presenteeism Score: number analyzed (Participants) | 96
  BUF-WPAI: Presenteeism Score | 0.50 [0.33 to 0.63]
  BUF-WPAI: Activity Impairment Score: number analyzed (Participants) | 150
  BUF-WPAI: Activity Impairment Score | 0.60 [0.48 to 0.69]
  BUF-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 150
  BUF-Generalize Anxiety Disorder-7 Score | 0.35 [0.20 to 0.48]
  SDT-IBDQ: IBDQ Total score: number analyzed (Participants) | 145
  SDT-IBDQ: IBDQ Total score | 0.37 [0.22 to 0.50]
  SDT-IBDQ: Bowel symptoms: number analyzed (Participants) | 145
  SDT-IBDQ: Bowel symptoms | 0.36 [0.21 to 0.49]
  SDT-IBDQ: Systemic symptoms: number analyzed (Participants) | 145
  SDT-IBDQ: Systemic symptoms | 0.34 [0.19 to 0.48]
  SDT-IBDQ: Emotional function: number analyzed (Participants) | 145
  SDT-IBDQ: Emotional function | 0.32 [0.16 to 0.46]
  SDT-IBDQ: Social function: number analyzed (Participants) | 145
  SDT-IBDQ: Social function | 0.34 [0.19 to 0.48]
  SDT-WPAI: UC Work Productivity Loss Score: number analyzed (Participants) | 97
  SDT-WPAI: UC Work Productivity Loss Score | -0.29 [-0.46 to -0.10]
  SDT-WPAI: UC Absenteeism Score: number analyzed (Participants) | 108
  SDT-WPAI: UC Absenteeism Score | -0.18 [-0.36 to 0.01]
  SDT-WPAI: UC Presenteeism Score: number analyzed (Participants) | 97
  SDT-WPAI: UC Presenteeism Score | -0.30 [-0.47 to -0.11]
  SDT-WPAI: UC Activity Impairment Score: number analyzed (Participants) | 152
  SDT-WPAI: UC Activity Impairment Score | -0.29 [-0.43 to -0.14]
  SDT-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 152
  SDT-Generalize Anxiety Disorder-7 Score | -0.26 [-0.40 to -0.11]
  SDT-APU for BU: number analyzed (Participants) | 155
  SDT-APU for BU | -0.37 [-0.49 to -0.22]
  APU-IBDQ: IBDQ Total score: number analyzed (Participants) | 143
  APU-IBDQ: IBDQ Total score | -0.51 [-0.62 to -0.38]
  APU-IBDQ: Bowel symptoms: number analyzed (Participants) | 143
  APU-IBDQ: Bowel symptoms | -0.46 [-0.58 to -0.32]
  APU-IBDQ: Systemic symptoms: number analyzed (Participants) | 143
  APU-IBDQ: Systemic symptoms | -0.43 [-0.56 to -0.29]
  APU-IBDQ: Emotional function: number analyzed (Participants) | 143
  APU-IBDQ: Emotional function | -0.45 [-0.57 to -0.30]
  APU-IBDQ: Social function: number analyzed (Participants) | 143
  APU-IBDQ: Social function | -0.54 [-0.64 to -0.41]
  APU-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 96
  APU-WPAI: Work Productivity Loss Score | 0.43 [0.25 to 0.58]
  APU-WPAI: Absenteeism Score: number analyzed (Participants) | 107
  APU-WPAI: Absenteeism Score | 0.22 [0.03 to 0.40]
  APU-WPAI: Presenteeism Score: number analyzed (Participants) | 96
  APU-WPAI: Presenteeism Score | 0.41 [0.22 to 0.56]
  APU-WPAI: Activity Impairment Score: number analyzed (Participants) | 151
  APU-WPAI: Activity Impairment Score | 0.48 [0.34 to 0.59]
  APU-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 151
  APU-Generalize Anxiety Disorder-7 Score | 0.25 [0.09 to 0.39]
  UNRS: PGR-S | 0.64 [0.54 to 0.72]
  UNRS: PGI-C: number analyzed (Participants) | 153
  UNRS: PGI-C | 0.45 [0.31 to 0.56]
  UNRS: Mayo SF | 0.35 [0.20 to 0.48]
  UNRS: Mayo RB | 0.21 [0.05 to 0.35]
  UNRS: Abdominal Pain NRS | 0.62 [0.51 to 0.70]
  UNRS: Fatigue NRS | 0.58 [0.47 to 0.67]
  UNRS: Nocturnal Stool | 0.49 [0.36 to 0.59]
  BUF: PGR-S | 0.65 [0.56 to 0.73]
  BUF: PGI-C: number analyzed (Participants) | 153
  BUF: PGI-C | 0.45 [0.31 to 0.56]
  BUF: Mayo SF | 0.53 [0.40 to 0.63]
  BUF: Mayo RB | 0.22 [0.07 to 0.36]
  BUF: Abdominal Pain NRS | 0.55 [0.43 to 0.65]
  BUF: Fatigue NRS | 0.49 [0.36 to 0.60]
  BUF: Nocturnal Stool | 0.62 [0.51 to 0.70]
  SDT: PGR-S | -0.44 [-0.56 to -0.31]
  SDT:Absolute SF | -0.30 [-0.43 to -0.15]
  SDT: Mayo SF | -0.28 [-0.41 to -0.13]
  SDT: Mayo RB | -0.22 [-0.36 to -0.07]
  SDT: Abdominal Pain NRS | -0.44 [-0.55 to -0.30]
  SDT: Fatigue NRS | -0.30 [-0.43 to -0.15]
  SDT: Nocturnal Stool | -0.33 [-0.46 to -0.19]
  SDT: PGI-C: number analyzed (Participants) | 153
  SDT: PGI-C | -0.29 [-0.43 to -0.14]
  APU: PGR-S: number analyzed (Participants) | 153
  APU: PGR-S | 0.39 [0.25 to 0.52]
  APU: PGI-C: number analyzed (Participants) | 151
  APU: PGI-C | 0.35 [0.20 to 0.48]
  APU: Mayo SF: number analyzed (Participants) | 154
  APU: Mayo SF | 0.44 [0.30 to 0.55]
  APU: Mayo RB: number analyzed (Participants) | 154
  APU: Mayo RB | 0.22 [0.06 to 0.36]
  APU: Abdominal Pain NRS: number analyzed (Participants) | 153
  APU: Abdominal Pain NRS | 0.23 [0.07 to 0.37]
  APU: Fatigue NRS: number analyzed (Participants) | 153
  APU: Fatigue NRS | 0.29 [0.14 to 0.43]
  APU: Nocturnal Stool: number analyzed (Participants) | 153
  APU: Nocturnal Stool | 0.50 [0.37 to 0.61]

11. Secondary Outcome: Correlation Between Change From Baseline in Urgency Numeric Rating Scale (UNRS), Baseline in Bowel Urgency Frequency (BUF), Stool Deferral Time (SDT) and Absorbent Product Use (APU) Measures, With QoL/Functional Outcome Measures and UC Symptom Measures
Description: This outcome evaluates correlations between change from baseline in UNRS, BUF, SDT, APU, and PROs related to quality of life (QoL), functional outcomes, and UC symptoms. QoL is assessed using the Inflammatory Bowel Disease Questionnaire (IBDQ), a 32-item patient-completed tool with four domains: bowel (score range 10-70), systemic (5-35), emotional (12-84), and social (5-35). Each item is rated on a 7-point Likert scale (1 = very severe problem, 7 = not a problem at all); The total IBDQ score is calculated by summing the scores from all four domains and total score range is 32-224 (Higher = better QoL). Functional outcomes measures: Work Productivity and Activity Impairment (WPAI) questionnaire (four scores derived: absenteeism, presenteeism, productivity loss, activity impairment; each score 0-100%, higher = greater impairment) and Generalized Anxiety Disorder-7 (GAD-7;total score range 0-21, higher = more severe anxiety)... (Continued below due to character constraint)
Time Frame: Baseline, Week 12 UC symptom measures:Patient Global Rating of Severity (PGR-S)(1-6),Patient Global Impression of Change (PGI-C)(1-7),Mayo SF/RB (0-3),Abdominal pain/fatigue NRS (0-10),nocturnal stool frequency; higher=worse severity for all measures.
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | 300 mg Mirikizumab
Number analyzed (Participants) | 160
Spearman Correlation Coefficient
  UNRS-IBDQ: IBDQ Total score: number analyzed (Participants) | 134
  UNRS-IBDQ: IBDQ Total score | -0.546 [-0.654 to -0.414]
  UNRS-IBDQ: Bowel symptoms: number analyzed (Participants) | 134
  UNRS-IBDQ: Bowel symptoms | -0.522 [-0.634 to -0.385]
  UNRS-IBDQ: Systemic symptoms: number analyzed (Participants) | 134
  UNRS-IBDQ: Systemic symptoms | -0.473 [-0.594 to -0.329]
  UNRS-IBDQ: Emotional function: number analyzed (Participants) | 134
  UNRS-IBDQ: Emotional function | -0.485 [-0.604 to -0.342]
  UNRS-IBDQ: Social function: number analyzed (Participants) | 134
  UNRS-IBDQ: Social function | -0.454 [-0.578 to -0.307]
  UNRS-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 72
  UNRS-WPAI: Work Productivity Loss Score | 0.488 [0.286 to 0.645]
  UNRS-WPAI: Absenteeism Score: number analyzed (Participants) | 98
  UNRS-WPAI: Absenteeism Score | 0.092 [-0.108 to 0.285]
  UNRS-WPAI: Presenteeism Score: number analyzed (Participants) | 72
  UNRS-WPAI: Presenteeism Score | 0.509 [0.312 to 0.661]
  UNRS-WPAI: Activity Impairment Score: number analyzed (Participants) | 145
  UNRS-WPAI: Activity Impairment Score | 0.451 [0.309 to 0.571]
  UNRS-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 145
  UNRS-Generalize Anxiety Disorder-7 Score | 0.179 [0.015 to 0.331]
  BUF-IBDQ: IBDQ Total score: number analyzed (Participants) | 134
  BUF-IBDQ: IBDQ Total score | -0.399 [-0.532 to -0.245]
  BUF-IBDQ: Bowel symptoms: number analyzed (Participants) | 134
  BUF-IBDQ: Bowel symptoms | -0.380 [-0.515 to -0.223]
  BUF-IBDQ: Systemic symptoms: number analyzed (Participants) | 134
  BUF-IBDQ: Systemic symptoms | -0.353 [-0.492 to -0.194]
  BUF-IBDQ: Emotional function: number analyzed (Participants) | 134
  BUF-IBDQ: Emotional function | -0.278 [-0.427 to -0.113]
  BUF-IBDQ: Social function: number analyzed (Participants) | 134
  BUF-IBDQ: Social function | -0.378 [-0.514 to -0.222]
  BUF-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 72
  BUF-WPAI: Work Productivity Loss Score | 0.275 [0.044 to 0.475]
  BUF-WPAI: Absenteeism Score: number analyzed (Participants) | 98
  BUF-WPAI: Absenteeism Score | 0.150 [-0.051 to 0.338]
  BUF-WPAI: Presenteeism Score: number analyzed (Participants) | 72
  BUF-WPAI: Presenteeism Score | 0.275 [0.045 to 0.475]
  BUF-WPAI: Activity Impairment Score: number analyzed (Participants) | 145
  BUF-WPAI: Activity Impairment Score | 0.356 [0.203 to 0.489]
  BUF-WPAI: Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 145
  BUF-WPAI: Generalize Anxiety Disorder-7 Score | 0.130 [-0.034 to 0.287]
  SDT-IBDQ: IBDQ Total score: number analyzed (Participants) | 136
  SDT-IBDQ: IBDQ Total score | 0.22 [0.05 to 0.38]
  SDT-IBDQ: Bowel symptoms: number analyzed (Participants) | 136
  SDT-IBDQ: Bowel symptoms | 0.26 [0.10 to 0.41]
  SDT-IBDQ: Systemic symptoms: number analyzed (Participants) | 136
  SDT-IBDQ: Systemic symptoms | 0.18 [0.01 to 0.34]
  SDT-IBDQ: Emotional function: number analyzed (Participants) | 136
  SDT-IBDQ: Emotional function | 0.16 [-0.01 to 0.32]
  SDT-IBDQ: Social function: number analyzed (Participants) | 136
  SDT-IBDQ: Social function | 0.15 [-0.02 to 0.31]
  SDT-WPAI: UC Work Productivity Loss Score: number analyzed (Participants) | 73
  SDT-WPAI: UC Work Productivity Loss Score | -0.14 [-0.36 to 0.09]
  SDT-WPAI: UC Absenteeism Score: number analyzed (Participants) | 99
  SDT-WPAI: UC Absenteeism Score | 0.03 [-0.17 to 0.22]
  SDT-WPAI: UC Presenteeism Score: number analyzed (Participants) | 73
  SDT-WPAI: UC Presenteeism Score | -0.17 [-0.38 to -0.06]
  SDT-WPAI: UC Activity Impairment Score: number analyzed (Participants) | 147
  SDT-WPAI: UC Activity Impairment Score | -0.17 [-0.32 to -0.00]
  SDT-Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 147
  SDT-Generalize Anxiety Disorder-7 Score | 0.03 [-0.14 to 0.19]
  SDT- APU for BU: number analyzed (Participants) | 152
  SDT- APU for BU | 0.07 [-0.09 to 0.23]
  APU-IBDQ: IBDQ Total score: number analyzed (Participants) | 135
  APU-IBDQ: IBDQ Total score | -0.290 [-0.436 to -0.126]
  APU-IBDQ: Bowel symptoms: number analyzed (Participants) | 135
  APU-IBDQ: Bowel symptoms | -0.240 [-0.392 to -0.073]
  APU-IBDQ: Systemic symptoms: number analyzed (Participants) | 135
  APU-IBDQ: Systemic symptoms | -0.160 [-0.319 to 0.010]
  APU-IBDQ: Emotional function: number analyzed (Participants) | 135
  APU-IBDQ: Emotional function | -0.258 [-0.409 to -0.093]
  APU-IBDQ: Social function: number analyzed (Participants) | 135
  APU-IBDQ: Social function | -0.321 [-0.464 to -0.160]
  APU-WPAI: Work Productivity Loss Score: number analyzed (Participants) | 72
  APU-WPAI: Work Productivity Loss Score | 0.040 [-0.194 to 0.269]
  APU-WPAI: Absenteeism Score: number analyzed (Participants) | 98
  APU-WPAI: Absenteeism Score | -0.031 [-0.228 to 0.169]
  APU-WPAI: Presenteeism Score: number analyzed (Participants) | 72
  APU-WPAI: Presenteeism Score | 0.030 [-0.204 to 0.259]
  APU-WPAI: Activity Impairment Score: number analyzed (Participants) | 146
  APU-WPAI: Activity Impairment Score | 0.153 [-0.010 to 0.308]
  APU-WPAI: Generalize Anxiety Disorder-7 Score: number analyzed (Participants) | 146
  APU-WPAI: Generalize Anxiety Disorder-7 Score | 0.139 [-0.025 to 0.294]
  UNRS: PGR-S | 0.672 [0.575 to 0.748]
  UNRS: Mayo SF | 0.478 [0.348 to 0.589]
  UNRS: Mayo RB | 0.368 [0.225 to 0.494]
  UNRS: Abdominal Pain NRS | 0.667 [0.570 to 0.744]
  UNRS: Fatigue NRS | 0.601 [0.491 to 0.691]
  UNRS: Nocturnal Stool | 0.191 [0.036 to 0.335]
  BUF: PGR-S | 0.502 [0.375 to 0.609]
  BUF: Mayo SF | 0.477 [0.346 to 0.587]
  BUF: Mayo RB | 0.351 [0.207 to 0.480]
  BUF: Abdominal Pain NRS | 0.399 [0.258 to 0.521]
  BUF: Fatigue NRS | 0.404 [0.264 to 0.525]
  BUF: Nocturnal Stool | 0.579 [0.464 to 0.672]
  SDT: PGR-S | -0.44 [-0.55 to -0.30]
  SDT: Absolute SF | -0.23 [-0.37 to -0.08]
  SDT: Mayo SF | -0.35 [-0.48 to -0.21]
  SDT: Mayo RB | -0.22 [-0.37 to -0.07]
  SDT: Abdominal Pain NRS | -0.39 [-0.52 to -0.25]
  SDT: Fatigue NRS | -0.30 [-0.43 to -0.15]
  SDT: Nocturnal Stool | -0.07 [-0.22 to 0.09]
  APU: PGR-S: number analyzed (Participants) | 150
  APU: PGR-S | 0.047 [-0.114 to 0.206]
  APU: Mayo SF: number analyzed (Participants) | 151
  APU: Mayo SF | 0.177 [0.018 to 0.327]
  APU: Mayo RB: number analyzed (Participants) | 151
  APU: Mayo RB | 0.120 [-0.041 to 0.274]
  APU: Abdominal Pain NRS: number analyzed (Participants) | 150
  APU: Abdominal Pain NRS | 0.168 [0.008 to 0.319]
  APU: Fatigue NRS: number analyzed (Participants) | 150
  APU: Fatigue NRS | 0.154 [-0.007 to 0.306]
  APU: Nocturnal Stool: number analyzed (Participants) | 150
  APU: Nocturnal Stool | 0.115 [-0.047 to 0.270]

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 12
Description: All enrolled participants who received at least one dose of study drug (regardless of whether the participant does not receive the correct treatment or otherwise does not follow the protocol)
Arm/Group | 300 mg Mirikizumab
All-Cause Mortality (participants affected / at risk) | 0/172
Serious Adverse Events (participants affected / at risk) | 5/172
Other Adverse Events (participants affected / at risk) | 53/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg Mirikizumab (N=172)
Any event (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Any event (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Any event (Infections and infestations) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1)
Any event (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Any event (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg Mirikizumab (N=172)
Any event (Blood and lymphatic system disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Any event (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (3)
Any event (Gastrointestinal disorders) | 10 (11)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 3 (4)
Any event (General disorders) | 12 (13)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Infusion site reaction (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Any event (Hepatobiliary disorders) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2)
Any event (Infections and infestations) | 11 (11)
Covid-19 (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (7)
Viral infection (Infections and infestations) | 2 (2)
Any event (Metabolism and nutrition disorders) | 6 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Any event (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Any event (Nervous system disorders) | 6 (7)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Any event (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Any event (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Any event (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05767021/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT05767021/SAP_001.pdf